CLINICAL TRIAL: NCT04880876
Title: A Phase 3, Long-term Safety Study of Oral Eluxadoline Administered to Pediatric Participants With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: A Study Evaluating Oral Eluxadoline Administered to Pediatric Participants With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3030-302-002
Record Dates: First submitted 2021-04-16; First posted 2021-05-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome with Diarrhea IBSD IBS-D Irritable Bowel Syndrome Pediatric
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — eluxadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Open Label 6-11 years of age: Eluxadoline 50mg (Experimental): Eluxadoline two 25mg tablets, oral administration, twice daily with food. Take at approximately the same time each day.
  Interventions: Drug: 25mg Eluxadoline
- Open Label 12-17 years of age: Eluxadoline 100 mg (Experimental): Eluxadoline one 100mg tablet, oral administration, twice daily with food. May use 25mg tablets to administer 100mg dose. Take at approximately the same time each day.
  Interventions: Drug: 25mg Eluxadoline; Drug: 100mg Eluxadoline
- Double Blind 6-11 years of age: Eluxadoline 25mg (Experimental): Blinding will be accomplished via administration of a constant number of oral tablets in each age group (6 to 11 years of age and 12 to 17 years of age) where all participants in an age group will receive the same total number of oral tablets at each administration. Phase 2 completers who choose to remain on double-blind eluxadoline and received placebo in the lead-in Phase 2 study 3030-202-002 will be assigned to double-blind eluxadoline 25 mg BID
  Interventions: Drug: 25mg Eluxadoline
- Double Blind 6-11 years of age: Eluxadoline 50mg (Experimental): Blinding will be accomplished via administration of a constant number of oral tablets in each age group (6 to 11 years of age and 12 to 17 years of age) where all participants in an age group will receive the same total number of oral tablets at each administration. Phase 2 completers who choose to remain on double-blind eluxadoline and received placebo in the lead-in Phase 2 study 3030-202-002 will be assigned to double-blind eluxadoline 25 mg BID
  Interventions: Drug: 25mg Eluxadoline
- Double Blind 12-17 years of age: Eluxadoline 25mg (Experimental): Blinding will be accomplished via administration of a constant number of oral tablets in each age group (6 to 11 years of age and 12 to 17 years of age) where all participants in an age group will receive the same total number of oral tablets at each administration. Phase 2 completers who choose to remain on double-blind eluxadoline and received placebo in the lead-in Phase 2 study 3030-202-002 will be assigned to double-blind eluxadoline 25 mg BID
  Interventions: Drug: 25mg Eluxadoline
- Double Blind 12-17 years of age: Eluxadoline 50mg (Experimental): Blinding will be accomplished via administration of a constant number of oral tablets in each age group (6 to 11 years of age and 12 to 17 years of age) where all participants in an age group will receive the same total number of oral tablets at each administration. Phase 2 completers who choose to remain on double-blind eluxadoline and received placebo in the lead-in Phase 2 study 3030-202-002 will be assigned to double-blind eluxadoline 25 mg BID
  Interventions: Drug: 25mg Eluxadoline
- Double Blind 12-17 years of age: Eluxadoline 100mg (Experimental): Blinding will be accomplished via administration of a constant number of oral tablets in each age group (6 to 11 years of age and 12 to 17 years of age) where all participants in an age group will receive the same total number of oral tablets at each administration. Phase 2 completers who choose to remain on double-blind eluxadoline and received placebo in the lead-in Phase 2 study 3030-202-002 will be assigned to double-blind eluxadoline 25 mg BID
  Interventions: Drug: 25mg Eluxadoline

INTERVENTIONS:
Drug: 25mg Eluxadoline — Oral Tablets
Drug: 100mg Eluxadoline — Oral Tablets
  Arms: Open Label 12-17 years of age: Eluxadoline 100 mg

SUMMARY:
This study will assess the long-term safety of oral Eluxadoline administered to pediatric participants with IBS-D who have completed study intervention in the Phase 2 study 3030-202-002 or the Phase 3 study 3030-303-002.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Male or female participants must be 6 to 17 years of age (inclusive)
* Participants must have completed study intervention in their lead-in study

Exclusion Criteria:

* Participant has an unresolved AE or a clinically significant finding on a physical examination, vital sign assessment, or neurological assessment along with an ECG or clinical laboratory tests (if results are available by the time of enrollment) that; in the opinion of the investigator, could represent a safety concern or a condition that would be exclusionary, could prevent the participant from performing any protocol assessments, or could confound study assessments.
* Participant has known allergies or hypersensitivity to opioids
* Female participants who are currently pregnant or nursing, or plan to become pregnant or nurse during the clinical study.
* Participant has no gallbladder, (ie, agenesis of the gallbladder or cholecystectomy).
* Participant has known or suspected biliary duct obstruction, or sphincter of Oddi disease or dysfunction
* Participant has a history of pancreatitis; structural diseases of the pancreas, known or suspected pancreatic duct obstruction
* Participant has a history of chronic or severe constipation, or sequelae from constipation, or known or suspected mechanical GI obstruction or pseudo obstruction
* Participant has renal impairment or an unstable hepatic, metabolic, or hematologic condition.
* Participant is a current regular alcohol drinker and/or binge drinker*, and/or has a history of alcoholism, alcohol abuse (eg, binge-drinking*), or alcohol addiction, and/or intends to consume alcohol during the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | 52 weeks
Percentage of Participants with Clinically Significant Laboratory Values (clinical chemistry, complete blood count, urinalysis) as assessed by the Investigator | 52 weeks
Percentage of Participants with Clinically Significant ECGs as assessed by the Investigator | 52 weeks
Percentage of Participants with Clinically Significant vital sign measurements as assessed by the Investigator | 52 weeks
Percentage of Participants with any new Physical examination abnormality or worsening of change from baseline | 52 weeks
Percentage of Participants with any new neurological abnormality post baseline or worsening of change from baseline | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- United States (6):
  - Kindred Medical Institute, LLC /ID# 227595, Corona, California
  - Valencia Medical & Research Center /ID# 246221, Miami, Florida
  - Florida Research Center, Inc. /ID# 227597, Miami, Florida
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 227600, Stockbridge, Georgia
  - IPS Research Company /ID# 227594, Oklahoma City, Oklahoma
  - Preferred Primary Care Physicians, Inc. /ID# 227596, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/